CLINICAL TRIAL: NCT05119777
Title: Prospective, Open Label, Post Marketing Study of the Safety and Effectiveness of HArmonyCa Injectable Gel for Mid-face Soft Tissue Augmentation
Brief Title: HArmonyCa Injectable Gel for Mid Face Soft Tissue Augmentation
Acronym: HArmonyCa EUMD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M21-787; 2021-A01899-32 (Other: AbbVie)
Record Dates: First submitted 2021-11-04; First posted 2021-11-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Soft Tissue Augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HArmonyCa Injectable Gel (Experimental): HArmonyCa injected at the discretion of the Treating Investigator (TI) to the midface for initial treatment and an optional touch-up treatment 14 days later
  Interventions: Device: HArmonyCa Injectable Gel

INTERVENTIONS:
Device: HArmonyCa Injectable Gel — Subdermal or deep dermal injection

SUMMARY:
Prospective, open label, post marketing study of the safety and effectiveness of HArmonyCa injectable gel for mid-face soft tissue augmentation

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 or older at the time of signing the ICF
* In general good health
* Participant seeking soft tissue augmentation in the mid face
* Has moderate or severe mid face volume deficit (Grade 5, 4, or 3 on the MFVDS) for each cheek on EI (Evaluating Investigator) live assessment (both cheeks must qualify but do not need to have the same score)
* Each cheek is amenable to achieving at least a 1-point improvement on the MFVDS with study intervention in the judgment of the EI (Evaluating Investigator)/TI (Treating Investigator)
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in the protocol
* Written informed consent from the participant has been obtained prior to any study-related procedures
* Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable
* Able, as assessed by the EI, and willing to follow study instructions (including compliance with the safety diary) and likely to complete all required study visits
* Fluent and literate in French

Exclusion Criteria:

* HArmonyCa is contraindicated:

  1. in patients with a known sensitivity to any of the product components.
  2. in patients suffering from skin disease or abnormal skin conditions.
  3. in patients suffering from an infection or inflammation (either acute or chronic) at or near the treatment site.
  4. in patients susceptible to keloid formation, hypertrophic scarring, or developing inflammatory skin conditions.
  5. in patients with impaired wound healing due to systemic disorders, medicinal drugs, or unhealthy or poorly-vascularized tissue.
  6. in patients suffering from prolonged bleeding or tissue healing due to medical conditions or medicinal drugs.
  7. in patients with a history of anaphylactic reactions and/or multiple severe allergies.
  8. in patients with a known sensitivity to steroids, or who are contraindicated to be treated with steroids.
  9. for injection into the glabellar or periocular areas.
  10. for injection into the lips and perioral region.
  11. for injection into regions containing foreign bodies.
  12. in patients presenting with herpes.
  13. in patients with autoimmune diseases.
  14. for injection into blood vessels and to highly vascularized areas.
  15. for injection into the epidermis or superficial dermis.
  16. in breastfeeding or pregnant women.
  17. in patients below the age of 18.
* Has experienced trauma to the face within 6 months before enrollment or has residual deficiencies, deformities, or scarring
* History of anaphylaxis or allergy to HA products, or Streptococcal protein
* Fat injection or permanent facial implants (eg, polymethylmethacrylate, silicone, polytetrafluoroethylene) anywhere in the face
* Semi-permanent soft-tissue filler treatment (eg, CaHA, poly-L-lactic acid) in the face within 36 months before enrollment
* Temporary dermal filler injections in the face within 24 months before enrollment
* Botulinum toxin treatment in the cheek area (including crow's feet, depressor anguli oris, jawline, platysma, etc.) within 6 months before enrollment
* Mesotherapy or cosmetic facial procedures in the face within 6 months before enrollment. Examples of mesotherapy or cosmetic facial procedures are face-lift, laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, moderate or greater depth chemical peel, or other ablative procedures.
* Changes in use of over-the-counter or prescription oral or topical, anti-wrinkle products in the face within 30 days before enrollment or planned changes during the study. Participants are not eligible for this study if they have begun using any new over-the-counter or prescription oral or topical, anti-wrinkle products in the face within 30 days before enrollment or are planning to begin using such products during the study. Participants who have been on a regimen of such products for at least 30 days are eligible for the study if they intend to continue their regimen throughout the study.
* Is on a regimen of anti-coagulation therapy (eg, warfarin, clopidogrel)
* Has received LASIK surgery or other surgical intervention on the eye within 3 months prior to enrollment or is planning such a procedure
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study
* Has tattoos, piercings, facial hair, or scars in the face that would interfere with the visualization of the face for the effectiveness assessment
* Has undergone a dental procedure within 6 weeks before treatment or plans to undergo a dental procedure (other than prophylaxis or dental fillings) during the course of the study
* Females who are pregnant, planning a pregnancy, or nursing.
* TI's discretion based on participant's safety and/or study integrity. The participant has a condition or is in a situation that, in the TI's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study.
* Directly or indirectly involved in the conduct and administration of this study. Directly or indirectly involved in the conduct and administration of this study as an investigator, sub-investigator, study coordinator, or other study staff member; employee of the sponsor; first degree family member, significant other, or relative residing with one of the above persons involved directly or indirectly in the study; or enrolled in the study at another clinical site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Responder status of achieving ≥ 1-grade improvement from baseline on Mid Face Volume Deficit Scale (MFVDS) based on EI's (Evaluating Investigator) live assessment at Month 1 | 1 Month
  The MFVDS is a validated, 6-point scale with grades of severe (5), significant (4), moderate (3), mild (2), minimal (1), and none (0)

SECONDARY OUTCOMES:
Responder status of achieving improved or much improved on Global Aesthetic Improvement Scale (GAIS) based on EI live assessment at Month 1 visit | 1 Month
  The GAIS is a validated, 5-point scale with grades of much improved (2), improved (1), no change (0), worse (-1), and much worse (-2)
Responder status of achieving improved or much improved on GAIS based on participant assessment at Month 1 visit | 1 Month
  The GAIS is a validated, 5-point scale with grades of much improved (2), improved (1), no change (0), worse (-1), and much worse (-2)
Change from baseline on FACE-Q Satisfaction with Cheeks specific questionnaire at Month 1 visit | 1 Month
  The FACE-Q is a validated 4-item Satisfaction with Cheeks questionnaire evaluated by the participant (very dissatisfied, somewhat dissatisfied, somewhat satisfied, very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (2):
- France (2):
  - Eurofins Dermscan Pharmascan /ID# 240921, Aix-en-Provence
  - Eurofins Pharmascan /ID# 240920, Lyon

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M21-787#additional-resources-section